CLINICAL TRIAL: NCT04337632
Title: Evaluation of the Sensitivity to Different Chemotherapy Regimens in Platinum-Partial Sensitive Recurrent Ovarian Cancer Based on 11 Gene Tests of Homologous Recombination Pathway
Brief Title: Evaluation of the Sensitivity to Different Chemotherapy Regimens in Platinum-Partial Sensitive Recurrent Ovarian Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Principal Investigator, JingWang, Professor, Hunan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016YFC1303703
Record Dates: First submitted 2020-03-26; First posted 2020-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — CP protocol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PP (Experimental): Doxorubicin Hydrochloride Liposome Injection 25mg/m2, carboplatin AUC 5, day 1, intravenous drip, repeated every three weeks.
  Interventions: Drug: Doxorubicin Hydrochloride Liposome Injection+carboplatin
- TP (Active Comparator): paclitaxel 175mg/m2, carboplatin AUC 5, day 1, intravenous infusion, repeated every three weeks.
  Interventions: Drug: paclitaxel +carboplatin

INTERVENTIONS:
Drug: Doxorubicin Hydrochloride Liposome Injection+carboplatin — Doxorubicin Hydrochloride Liposome Injection 25mg/m2, carboplatin AUC 5, first day, intravenous drip, repeated every three weeks.
  Other Names: PP
  Arms: PP
Drug: paclitaxel +carboplatin — paclitaxel 175mg/m2, carboplatin AUC 5, day 1, intravenous infusion, repeated every three weeks.
  Other Names: TP
  Arms: TP

SUMMARY:
Multicenter, prospective, randomized studies.Evaluation of the sensitivity to different chemotherapy regimens in platinum-partial sensitive recurrent ovarian cancer based on 11 gene tests of homologous recombination pathway.

DETAILED DESCRIPTION:
Patients meeting the following inclusion criteria were randomly divided into two groups in a 1:1 ratio: paclitaxel/platinum chemotherapy group (TP) and Doxorubicin Hydrochloride Liposome Injection/platinum chemotherapy group (PP) (the specific chemotherapy regimens are as follows.Chemotherapy to tumor progression or adverse reactions can not be tolerated, effective chemotherapy patients with a maximum of 6 cycles of chemotherapy.The primary endpoint was progression-free survival (PFS), and the secondary endpoints were safety and overall survival.Also USES the next-generation sequencing (NGS) method to detect patients with recurrence after tumor tissues (including chest, ascites, homologous recombination pathway in the tumor tissue and peripheral blood ctDNA 11 genetic mutations, rearrangement, and so on and so forth, whether patients with analysing the homologous recombination pathways for paclitaxel/platinum chemotherapy or Doxorubicin Hydrochloride Liposome Injection/platinum chemotherapy has different sensitivity.

ELIGIBILITY:
Inclusion Criteria:

1. age: 18-75 years old
2. PS score: ECOG 0 ~ 2
3. histopathologically confirmed primary high-grade serous adenocarcinoma or high-grade endometrioid adenocarcinoma of the ovary, fallopian tube or peritoneum;
4. the time interval between this recurrence and the last chemotherapy was 6-12 months;
5. evaluate the ability of bone marrow, liver, kidney, heart and other important organ functions to withstand chemotherapy;
6. expected survival over 3 months;
7. sign the informed consent.

Exclusion Criteria:

1. brain metastasis or the presence of symptoms caused by brain metastasis;
2. serious complications;
3. acute inflammatory reaction;
4. other tumors;
5. a history of allergy to paclitaxel or polyropyridone liposomes;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
PFS（Progression-Free-Survival) | up to 24months
  From the date of randomization to the time of tumor progression

SECONDARY OUTCOMES:
OS(Overall survival) | up to 36months
  Time from random day to death (month)
ORR( Objective response rate) | up to 12 months
  the percentage of patients whose tumors shrink a certain amount and stay that way for a certain amount of time

CONTACTS AND LOCATIONS:
Overall Officials: Jing Wang, MD., Study Chair — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China